CLINICAL TRIAL: NCT02265107
Title: Effects of Exercise Training on Vascular Endothelial Function of Patients Submitted to Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande (FURG) (Other)
Responsible Party: Principal Investigator, Priscila Aikawa, Priscila Aikawa PhD, Universidade Federal do Rio Grande (FURG)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRC-FMD-2014
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Vasodilation
Keywords: endothelial function; physical training; exercise; coronary artery bypass
MeSH Terms: conditions — Aneurysm; Motor Activity | interventions — Exercise; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- cardiac rehabilitation (Experimental): We invited all consecutive patients submitted to CABG alone at Cardiologic Hospital Doctor Pedro Bertoni of the Associação de Caridade Santa Casa do Rio Grande in the period of October, 2011 until October, 2012, who resided in the city of the Rio Grande (RS/Brazil), to participate of the exercise training (ET). All patients were evaluated by cardiologist, and were ranked in Functional Classification of New York Heart Association (NYHA) such class I and II. Initially, twenty-four patients accepted and start to participate of ET, but only nine patients completed the program until the end.
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — The program of exercise training (ET) was employed for 6 consecutive months with 3 sessions per week. The training of physical activity consisted of a combination of aerobic and resistance exercises for upper and lower limbs. Each session included: (1) 5-minute warm-up, (2) 30 minutes of aerobic exercise (performed in treadmills and stationary bikes); (3) 20 minutes of resistance exercises with dumbbells for upper limbs and ankle support for lower limbs (exercises preformed in diagonals) that consisted of 6 sets of 10 resistance exercises repeated for upper limbs, and the same number of sets for lower limbs; and (4) 5-minute cool-down, totaling ninety minutes of session per day (90min/day) and, two hundred and seventy minutes per week (270min/week).
  Other Names: cardiac rehabilitation

SUMMARY:
Objective: To observe the effects of exercise training on vascular endothelial function in patients undergoing coronary artery bypass graft (CABG) alone in phase III after six months of Cardiac rehabilitation programs (CRP).

Methods: the investigators contacted all patients undergoing CABG alone in period of 1 year to participate in a CRP with duration of six months with three weekly sessions of 1 and half hour of the duration. All patients underwent biochemical blood tests, muscle strength testing of one repetition maximum (1-RM test) for upper and lower limbs, 6-minute walk test (6MWT), and evaluation of endothelial function (using flow-mediated vasodilation).

DETAILED DESCRIPTION:
Introduction The cardiac rehabilitation optimizes a cardiac patient's physical, psychological, and social functioning, in addition to stabilizing, slowing, or even reversing the progression of the underlying atherosclerotic processes, thereby reducing morbidity and mortality. Patients who recently had had a myocardial infarction; or had undergone coronary artery bypass graft; or who had undergone percutaneous coronary interventions; or who are heart transplantation candidates or recipients; or have stable chronic heart failure, peripheral arterial disease with claudication, or other forms of CVD are candidates eligible for cardiac rehabilitation services ( , ).

Recently, studies randomized clinical trials have reported the efficacy of the exercise training (ET) independently of format of exercise: aerobic, resistance, or combined exercise training in patients with coronary artery disease ( , ) and, others studies investigated the effects of ET on vascular endothelial function in patients with stable coronary artery disease ( ), ischemic heart disease ( ), recent myocardial infarction (4), and chronic heart failure (3, , ). ET is associated with an improvement in endothelial function, oxidative stress, and inflammation. Furthermore, the ET promotes beneficial effects on cardiovascular outcomes and decreases hospitalizations.

Arterial endothelium function evaluated by flow-mediated vasodilation (FMD) is a predictor of long-term adverse cardiovascular outcomes in healthy subjects ( ). Vascular endothelial dysfunction is an independent risk factor for cardiovascular events and provides important prognostic data in addition to the more traditional risk factors ( ). Endothelial dysfunction plays an important role in patients with coronary atherosclerosis (both acute and chronic myocardial ischemia) and heart failure (3,5, ). Therefore, we aim to investigate the effect of combined exercise training on vascular endothelial function in sedentary patients submitted to coronary artery bypass graft (CABG) in late phase.

Methods The protocol was approved by the local ethics committee of Associação de Caridade Santa Casa do Rio Grande Hospital, Rio Grande/RS - Brazil, under the protocol number 003/2013. This study was non-randomized clinical trial. The written informed consent was obtained from all patients before of the onset of ET. The investigators invited all consecutive patients submitted to CABG alone at Cardiologic Hospital Doctor Pedro Bertoni of the Associação de Caridade Santa Casa do Rio Grande in the period of October, 2011 until October, 2012, who resided in the city of the Rio Grande (RS/Brazil), to participate of the ET. The investigators excluded the patients that performed others cardiologic procedures with the CABG. All patients were evaluated by cardiologist, and were ranked in Functional Classification of New York Heart Association (NYHA) such class I and II. Initially, twenty-four patients accepted and start to participate of ET, but only nine patients completed the program until the end.

The program of exercise training (ET) was employed for 6 consecutive months with 3 sessions per week. The training of physical activity consisted of a combination of aerobic and resistance exercises for upper and lower limbs. Each session included: (1) 5-minute warm-up, (2) 30 minutes of aerobic exercise (performed in treadmills and stationary bikes); (3) 20 minutes of resistance exercises with dumbbells for upper limbs and ankle support for lower limbs (exercises preformed in diagonals) that consisted of 6 sets of 10 resistance exercises repeated for upper limbs, and the same number of sets for lower limbs; and (4) 5-minute cool-down, totaling ninety minutes of session per day (90min/day) and, two hundred and seventy minutes per week (270min/week) ( ). Initialy, in aerobic exercises, the maximal HR to be achieved was established between 30-40% of HR at rest and, the aerobic exercise was limited by symptoms reported by patients. The initial weight of the dumbbells and ankle were established between 30-40% of one-repetition maximum test (1-RM test) and, gradually increased according to the symptoms reported by patients, without compensation of the trunk to perform the exercises, no history of muscle pain, and no muscle fatigue to complete all sessions. Heart rate (HR), respiratory rate (RR), saturation pulse of oxygen, and blood pressure were measured at the beginning, middle and end of each session. The intensity and the velocity of the exercise program were progressively increased.

The baseline assessment was performed before the beginning of ET and, consisted of: blood chemistry (glycemia, insulin, glycohemoglobin, total-, high-, and low-density lipoprotein cholesterol, triglycerides); body mass index; strength of upper and lower limbs by 1-RM test of biceps brachialis and quadriceps, respectively; evaluation of functional capacity and; evaluation of vascular endothelial function.

Cholesterol, triglycerides, high-density lipoproteins (HDLc) and, glucose urea were measured using LAB TEST commercial kits (Lagoa Santa, MG, Brazil) and analyzed in LAB MAX 240® (Tokyo, Japan) equipment. The low density lipoproteins (LDLc) was calculated by Friedewald's formula. Glucose levels were measured by Trinder assay (calorimetry) in the equipment LAB MAX 240® (Tokyo, Japan). The insulin was assessed by chemiluminescence method using the Immulite® DPC equipment (Diagnostic Products Corporation - DPC, Los Angeles, CA, USA). The glycosylated hemoglobin (HbA1c) was determined by enzymatic method using the equipment LAB MAX 240® (Tokyo, Japan).

The 6-minutes walking test (6MWT) is used to assess the functional capacity of the individual, which is extremely important to evaluate tolerance and exercise capacities for the evaluation clinical and prognosis of patients with cardiovascular and pulmonary diseases ( , ). The 6MWT was performed on the first day in a linear corridor with 40 meters of length, and the researcher performed the test giving verbal commands to the patient, which should be done the best speed supported by him, and the researcher asked to the patient what their physical sensations. Data were collected before, at 3 minutes and at the end of the test for respiratory rate (RR), heart rate (HR), saturation pulse in portable pulse oximeter (Nonin®, model 9500, Plymouth, USA), and blood pressure systemic.

Flow-mediated vasodilation (FMD) was measured to evaluating arterial endothelium-dependent vasodilation using a high-resolution vascular ultrasound (Logiq P6, GE Healtcare, GE Ultrasound Korea Ltda.) according to American Heart Association Guideline ( ) with adjustments ( , ). Settings of depth and gain imaging were kept constant throughout the study. Briefly, changing in brachial artery diameter after 60 s of reactive hyperemia, after deflation of a cuff placed around the upper arm and inflated to 50 mmHg above the systolic blood pressure during five min, was compared with a baseline measurement. To evaluate basal blood flow and flow immediately after cuff release obtained no later than 15 s after cuff deflation we used a pulsed-wave Doppler velocity signals (assessed using Doppler bean-vessel angle ≤60º). The increased diameter after a sublingual nitroglycerin spray (0.4 mg) was used as a measurement of endothelium-independent vasodilation. The vessel diameter responses to reactive hyperemia and to nitroglycerin were expressed as the percentage changing relative to diameter immediately before cuff inflation and to diameter immediately before drug administration. Measurements of brachial artery diameter were accomplished off line by two evaluators using a semiautomatic quantitative analysis system after interventions. The second evaluator performing measures was blind to first evaluator's measures. Differences larger than 0.01 mm between assessors (mean vessel diameter) repeated were repeated. All data were measured twice, and final values were present as mean.

A nutritional counseling was performed, in wich the patients were instructed to avoid consumption of saturated fat and high-calorie foodstuff, to intake of dietary fiber, to maintain good hydration and to implement a fractionation of meals throughout the day, besides to receive instructions of food preparation, according to "I Diretriz sobre o Consumo de Gorduras e Saúde Cardiovascular" in "Arquivos Brasileiros de Cardiologia" of the "Sociedade Brasileira de Cardiologia" ( ).

All tests were repeated after 6 months, and the results were compared to baseline tests. The training program was stopped at this point.

The data are presented as the means ± SD. Distribution of variables was tested by Shapiro Wilk normality test. Baseline values were compared to values after 6 months of training program by use paired t-test. A value of P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* resided in the city of the Rio Grande (RS/Brazil);
* age over 18 years-old;
* evaluation and medical authorization.

Exclusion Criteria:

* the patients that performed others cardiologic procedures with the Coronary Artery Bypass Graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial function | after 6 months

OTHER OUTCOMES:
6-minute walk test | 6 months
  The 6-minutes walking test (6MWT) is used to assess the functional capacity of the individual

CONTACTS AND LOCATIONS:
Locations (1):
- Priscila Aikawa, Rio Grande, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] Vuckovic KM, Piano MR, Phillips SA. Effects of exercise interventions on peripheral vascular endothelial vasoreactivity in patients with heart failure with reduced ejection fraction. Heart Lung Circ. 2013 May;22(5):328-40. doi: 10.1016/j.hlc.2012.12.006. Epub 2013 Jan 20. PMID 23340198
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Luk TH, Dai YL, Siu CW, Yiu KH, Chan HT, Lee SW, Li SW, Fong B, Wong WK, Tam S, Lau CP, Tse HF. Effect of exercise training on vascular endothelial function in patients with stable coronary artery disease: a randomized controlled trial. Eur J Prev Cardiol. 2012 Aug;19(4):830-9. doi: 10.1177/1741826711415679. Epub 2011 Jul 1. PMID 21724681
- [Background] Morikawa Y, Mizuno Y, Harada E, Katoh D, Kashiwagi Y, Morita S, Yoshimura M, Uemura S, Saito Y, Yasue H. Aerobic interval exercise training in the afternoon reduces attacks of coronary spastic angina in conjunction with improvement in endothelial function, oxidative stress, and inflammation. Coron Artery Dis. 2013 May;24(3):177-82. doi: 10.1097/MCA.0b013e32835cbef5. PMID 23249633
- [Background] Anagnostakou V, Chatzimichail K, Dimopoulos S, Karatzanos E, Papazachou O, Tasoulis A, Anastasiou-Nana M, Roussos C, Nanas S. Effects of interval cycle training with or without strength training on vascular reactivity in heart failure patients. J Card Fail. 2011 Jul;17(7):585-91. doi: 10.1016/j.cardfail.2011.02.009. Epub 2011 Apr 22. PMID 21703531
- [Background] Credeur DP, Mariappan N, Francis J, Thomas D, Moraes D, Welsch MA. Vasoreactivity before and after handgrip training in chronic heart failure patients. Atherosclerosis. 2012 Nov;225(1):154-9. doi: 10.1016/j.atherosclerosis.2012.08.013. Epub 2012 Sep 16. PMID 23010159
- [Background] Shechter M, Shechter A, Koren-Morag N, Feinberg MS, Hiersch L. Usefulness of brachial artery flow-mediated dilation to predict long-term cardiovascular events in subjects without heart disease. Am J Cardiol. 2014 Jan 1;113(1):162-7. doi: 10.1016/j.amjcard.2013.08.051. Epub 2013 Oct 5. PMID 24169007
- [Background] Lerman A, Zeiher AM. Endothelial function: cardiac events. Circulation. 2005 Jan 25;111(3):363-8. doi: 10.1161/01.CIR.0000153339.27064.14. No abstract available. PMID 15668353
- [Background] Fiorina C, Vizzardi E, Lorusso R, Maggio M, De Cicco G, Nodari S, Faggiano P, Dei Cas L. The 6-min walking test early after cardiac surgery. Reference values and the effects of rehabilitation programme. Eur J Cardiothorac Surg. 2007 Nov;32(5):724-9. doi: 10.1016/j.ejcts.2007.08.013. Epub 2007 Sep 18. PMID 17881241
- [Background] Signori LU, Quadros AS, Sbruzzi G, Dipp T, Lopes RD, Schaan BD. Endothelial function in patients with slow coronary flow and normal coronary angiography. Clinics (Sao Paulo). 2012;67(6):677-80. doi: 10.6061/clinics/2012(06)22. No abstract available. PMID 22760911
- [Background] Lee KW, Blann AD, Jolly K, Lip GY; BRUM Investigators. Plasma haemostatic markers, endothelial function and ambulatory blood pressure changes with home versus hospital cardiac rehabilitation: the Birmingham Rehabilitation Uptake Maximisation Study. Heart. 2006 Dec;92(12):1732-8. doi: 10.1136/hrt.2006.092163. Epub 2006 Jun 28. PMID 16807272
- [Background] Hambrecht R, Wolf A, Gielen S, Linke A, Hofer J, Erbs S, Schoene N, Schuler G. Effect of exercise on coronary endothelial function in patients with coronary artery disease. N Engl J Med. 2000 Feb 17;342(7):454-60. doi: 10.1056/NEJM200002173420702. PMID 10675425
- [Background] Gokce N, Vita JA, Bader DS, Sherman DL, Hunter LM, Holbrook M, O'Malley C, Keaney JF Jr, Balady GJ. Effect of exercise on upper and lower extremity endothelial function in patients with coronary artery disease. Am J Cardiol. 2002 Jul 15;90(2):124-7. doi: 10.1016/s0002-9149(02)02433-5. PMID 12106840
- [Background] Edwards DG, Schofield RS, Lennon SL, Pierce GL, Nichols WW, Braith RW. Effect of exercise training on endothelial function in men with coronary artery disease. Am J Cardiol. 2004 Mar 1;93(5):617-20. doi: 10.1016/j.amjcard.2003.11.032. PMID 14996592
- [Background] Ades PA. Cardiac rehabilitation and secondary prevention of coronary heart disease. N Engl J Med. 2001 Sep 20;345(12):892-902. doi: 10.1056/NEJMra001529. No abstract available. PMID 11565523
- [Background] Opasich C, De Feo S, Pinna GD, Furgi G, Pedretti R, Scrutinio D, Tramarin R. Distance walked in the 6-minute test soon after cardiac surgery: toward an efficient use in the individual patient. Chest. 2004 Dec;126(6):1796-801. doi: 10.1378/chest.126.6.1796. PMID 15596676
- [Background] Opasich C, Pinna GD, Mazza A, Febo O, Riccardi PG, Capomolla S, Cobelli F, Tavazzi L. Reproducibility of the six-minute walking test in patients with chronic congestive heart failure: practical implications. Am J Cardiol. 1998 Jun 15;81(12):1497-500. doi: 10.1016/s0002-9149(98)00218-5. PMID 9645905
- [Background] Lee DH, Buth KJ, Martin BJ, Yip AM, Hirsch GM. Frail patients are at increased risk for mortality and prolonged institutional care after cardiac surgery. Circulation. 2010 Mar 2;121(8):973-8. doi: 10.1161/CIRCULATIONAHA.108.841437. Epub 2010 Feb 16. PMID 20159833
- [Background] Kim C, Kim BO, Lim KB, Kim YJ, Park YB. The Effect of Power-walking in Phase 2 Cardiac Rehabilitation Program. Ann Rehabil Med. 2012 Feb;36(1):133-40. doi: 10.5535/arm.2012.36.1.133. Epub 2012 Feb 29. PMID 22506246
- [Background] Pavy B, Caillon M. [Effects of a cardiac rehabilitation programme in coronary patient according to age]. Ann Cardiol Angeiol (Paris). 2012 Nov;61(5):338-44. doi: 10.1016/j.ancard.2012.08.038. Epub 2012 Aug 30. French. PMID 23021239
- See also: Additional reference — http://circ.ahajournals.org/content/105/5/546.full
- See also: Additional reference — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1517-86922014000100055
- See also: Additional reference — http://www.scielo.br/scielo.php?script=sci_nlinks&ref=000145&pid=S0103-0582201200030001900034&lng=pt
- See also: Additional reference — http://www.physiomics.eu/media/37024/am_j_physiol_heart_circ_physiol_300_h2_h12__2011.pdf
- See also: Additional reference — http://publicacoes.cardiol.br/consenso/2013/Diretriz_Gorduras.pdf
- See also: Additional reference — http://bmjopen.bmj.com/content/4/5/e005268.full